CLINICAL TRIAL: NCT03548753
Title: Functional and Anatomical Testing in Intermediate Risk Chest Pain Patients With Severe Coronary Calcium Score
Brief Title: Use of FFR-CT in Stable Intermediate Chest Pain Patients With Severe Coronary Calcium Score
Acronym: FACC
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Hans Mickley, Professor (chair), MD, Odense University Hospital
Other Study IDs: HM19501968
Record Dates: First submitted 2018-05-22; First posted 2018-06-07 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Observational
Keywords: Angina; Chest pain; Diagnostic tests
MeSH Terms: conditions — Angina Pectoris; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Agatston score > 399: 1. Coronary computed tomography angiography with FFR-CT
  2. Invasive coronary angiography with FFR

SUMMARY:
A prospective, blinded multicenter study for evaluation of chest pain patients with severe coronary calcium (Agatston score > 399). The objective is to evaluate if an initial non-invasive strategy with coronary computed tomography angiography (CCTA) including functional flow reserve derived from CCTA (FFR-CT) is as effective as invasive coronary angiography (ICA) including functional flow reserve (FFR) for the detection and exclusion of obstructive coronary artery disease (CAD). Study hypothesis: initial non-invasive anatomic and functional testing is non-inferior to an invasive anatomic and functional testing strategy.

DETAILED DESCRIPTION:
Prospective, blinded multicenter study evaluating the diagnostic performance of coronary computed tomography angiography (CCTA) including functional flow reserve derived from CCTA (FFR-CT) for the detection and exclusion of significant obstructive coronary artery disease (CAD). The reference standard vil be invasive coronary angiography (ICA) including functional flow reserve (FFR). Patients referred for elective CCTA because of suspected stable CAD are considered. If the initial routine non-enhanced CT scan shows an Agatston score > 399, the patient is eligible for study inclusion. Four sites in the region of Southern Denmark will participate (Odense University Hospital, Svendborg Hospital, Vejle Hospital and Esbjerg Hospital). A total of 278 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* An estimated likelihood for the presence of significant CAD between 15% and 85%
* Clinical stable patients with symptoms of suspected CAD referred for CTTA
* Initial routine non-enhanced CT scan shows an Agatston score >399
* Written informed consent
* Accept to undergo elective invasive coronary angiography (ICA) within 90 days

Exclusion Criteria:

* Known prior myocardial infarction
* Prior percutaneous coronary intervention (PCI)
* Prior coronary artery bypass surgery (CABG)
* Pacemaker or internal defibrillator lead implantation
* Prosthetic heart valve
* Atrial fibrillation
* Renal Insufficiency (<40 mL/min)
* Known anaphylactic reaction to iodinated contrast
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Clinical stable outpatients with symptoms of suspected coronary artery disease (CAD) referred for coronary computed tomography angiography (CCTA) as first-line noninvasive diagnostic test at one of the four participating centers are eligible for study inclusion, if the initial routine non-enhanced CT scan shows an Agatston score > 399.
Sampling Method: Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Per-patient diagnostic accuracy of functional flow reserve (FFR-CT) derived from standard coronary computed tomography angiography (CCTA) compared to invasive coronary angiography (ICA) including functional flow ratio (FFR) | Comparison of the noninvasive and invasive diagnostic modalities is performed at least 90 days after enrollment of each of the included patients
  The primary outcome measure is the per-patient diagnostic accuracy of functional flow reserve (FFR-CT) derived from standard coronary computed tomography angiography (CCTA) compared to invasive coronary angiography (ICA) including functional flow ratio (FFR), which is considered the gold standard in the detection or exclusion of obstructive coronary artery disease (CAD)

SECONDARY OUTCOMES:
Invasive coronary angiography (ICA) including functional flow ratio (FFR) without obstructive coronary artery disease | 90 days after inclusion
  Percentage of patients with invasive coronary angiography (ICA) including functional flow reserve (FFR) measurement without evidence of obstructive coronary artery disease
Coronary revascularization procedures | 90 day after inclusion
  Percentage of coronary revascularization procedures (PCI and CABG) in patients with reduced FFR-CT vs. patients with normal FFR-CT
Other clinical endpoints | 90 days after inclusion
  Percentage of patients with the composite endpoint of all-cause mortality or myocardial infarction or unstable angina hospitalization
Major complications from diagnostic invasive diagnostic procedures | Within 72 hours after invasive procedure
  Percentage of patients with major complications following invasive coronary angiography (ICA) including fractional flow reserve (FFR) measurement
Per-patient and per-vessel diagnostic performance of FFR-CT by means of accuracy, sensitivity, specificity, positive predictive value, and negative predictive value | At least 90 days after patient inclusion
  Assessing per-patient and per-vessel diagnostic performance of FFR-CT by means of accuracy, sensitivity, specificity, positive predictive value, and negative predictive value
Per-vessel correlation of FFR-CT numerical value with the FFR numerical value in patients undergoing FFR | At least 90 days after patient inclusion
  The per-vessel correlation of FFRCT numerical value with the FFR numerical value in patients undergoing FFR
The diagnostic accuracy of FFR-CT in subgroups of patients with high calcium score vs. patients with very high calcium score | At least 90 days after patient inclusion
  Comparison of the diagnostic accuracy of FFR-CT in subgroups of patients with high calcium score (Agatston score 400-999) vs patients with very high calcium score (Agatston score ≥ 999)
Costs and resource use. | 90 days after inclusion
  Estimating the total costs of potentially unnecessary invasive coronary angiographies with functional flow ratio measurements

CONTACTS AND LOCATIONS:
Overall Officials: Hans Mickley, MD, Study Chair — Professor, MD, DMSc
Locations (1):
- Odense University Hospital, Odense, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu MT, Ferencik M, Roberts RS, Lee KL, Ivanov A, Adami E, Mark DB, Jaffer FA, Leipsic JA, Douglas PS, Hoffmann U. Noninvasive FFR Derived From Coronary CT Angiography: Management and Outcomes in the PROMISE Trial. JACC Cardiovasc Imaging. 2017 Nov;10(11):1350-1358. doi: 10.1016/j.jcmg.2016.11.024. Epub 2017 Apr 12. PMID 28412436
- [Background] Patel MR, Dai D, Hernandez AF, Douglas PS, Messenger J, Garratt KN, Maddox TM, Peterson ED, Roe MT. Prevalence and predictors of nonobstructive coronary artery disease identified with coronary angiography in contemporary clinical practice. Am Heart J. 2014 Jun;167(6):846-52.e2. doi: 10.1016/j.ahj.2014.03.001. Epub 2014 Mar 14. PMID 24890534
- [Background] Yan RT, Miller JM, Rochitte CE, Dewey M, Niinuma H, Clouse ME, Vavere AL, Brinker J, Lima JA, Arbab-Zadeh A. Predictors of inaccurate coronary arterial stenosis assessment by CT angiography. JACC Cardiovasc Imaging. 2013 Sep;6(9):963-72. doi: 10.1016/j.jcmg.2013.02.011. Epub 2013 Aug 8. PMID 23932641
- [Background] Kruk M, Noll D, Achenbach S, Mintz GS, Pregowski J, Kaczmarska E, Kryczka K, Pracon R, Dzielinska Z, Sleszycka J, Witkowski A, Demkow M, Ruzyllo W, Kepka C. Impact of coronary artery calcium characteristics on accuracy of CT angiography. JACC Cardiovasc Imaging. 2014 Jan;7(1):49-58. doi: 10.1016/j.jcmg.2013.07.013. Epub 2013 Nov 27. PMID 24290567
- [Background] Ong TK, Chin SP, Liew CK, Chan WL, Seyfarth MT, Liew HB, Rapaee A, Fong YY, Ang CK, Sim KH. Accuracy of 64-row multidetector computed tomography in detecting coronary artery disease in 134 symptomatic patients: influence of calcification. Am Heart J. 2006 Jun;151(6):1323.e1-6. doi: 10.1016/j.ahj.2005.12.027. PMID 16781246
- [Background] Koo BK, Erglis A, Doh JH, Daniels DV, Jegere S, Kim HS, Dunning A, DeFrance T, Lansky A, Leipsic J, Min JK. Diagnosis of ischemia-causing coronary stenoses by noninvasive fractional flow reserve computed from coronary computed tomographic angiograms. Results from the prospective multicenter DISCOVER-FLOW (Diagnosis of Ischemia-Causing Stenoses Obtained Via Noninvasive Fractional Flow Reserve) study. J Am Coll Cardiol. 2011 Nov 1;58(19):1989-97. doi: 10.1016/j.jacc.2011.06.066. PMID 22032711
- [Background] Norgaard BL, Leipsic J, Gaur S, Seneviratne S, Ko BS, Ito H, Jensen JM, Mauri L, De Bruyne B, Bezerra H, Osawa K, Marwan M, Naber C, Erglis A, Park SJ, Christiansen EH, Kaltoft A, Lassen JF, Botker HE, Achenbach S; NXT Trial Study Group. Diagnostic performance of noninvasive fractional flow reserve derived from coronary computed tomography angiography in suspected coronary artery disease: the NXT trial (Analysis of Coronary Blood Flow Using CT Angiography: Next Steps). J Am Coll Cardiol. 2014 Apr 1;63(12):1145-1155. doi: 10.1016/j.jacc.2013.11.043. Epub 2014 Jan 30. PMID 24486266
- [Background] Norgaard BL, Gaur S, Leipsic J, Ito H, Miyoshi T, Park SJ, Zvaigzne L, Tzemos N, Jensen JM, Hansson N, Ko B, Bezerra H, Christiansen EH, Kaltoft A, Lassen JF, Botker HE, Achenbach S. Influence of Coronary Calcification on the Diagnostic Performance of CT Angiography Derived FFR in Coronary Artery Disease: A Substudy of the NXT Trial. JACC Cardiovasc Imaging. 2015 Sep;8(9):1045-1055. doi: 10.1016/j.jcmg.2015.06.003. Epub 2015 Aug 19. PMID 26298072
- [Background] Hecht HS. Coronary artery calcium scanning: past, present, and future. JACC Cardiovasc Imaging. 2015 May;8(5):579-596. doi: 10.1016/j.jcmg.2015.02.006. PMID 25937196
- [Background] Douglas PS, Hoffmann U, Lee KL, Mark DB, Al-Khalidi HR, Anstrom K, Dolor RJ, Kosinski A, Krucoff MW, Mudrick DW, Patel MR, Picard MH, Udelson JE, Velazquez EJ, Cooper L; PROMISE investigators. PROspective Multicenter Imaging Study for Evaluation of chest pain: rationale and design of the PROMISE trial. Am Heart J. 2014 Jun;167(6):796-803.e1. doi: 10.1016/j.ahj.2014.03.003. Epub 2014 Mar 18. PMID 24890527
- [Derived] Mickley H, Veien KT, Gerke O, Lambrechtsen J, Rohold A, Steffensen FH, Husic M, Akkan D, Busk M, Jessen LB, Jensen LO, Diederichsen A, Ovrehus KA. Diagnostic and Clinical Value of FFRCT in Stable Chest Pain Patients With Extensive Coronary Calcification: The FACC Study. JACC Cardiovasc Imaging. 2022 Jun;15(6):1046-1058. doi: 10.1016/j.jcmg.2021.12.010. Epub 2022 Feb 16. PMID 35680213